CLINICAL TRIAL: NCT03763929
Title: Double-Blind, Randomized, Placebo-Controlled, Phase 2 Study of Efficacy and Safety of Trans Sodium Crocetinate (TSC) Administered Onboard Emergency Vehicles for Treatment of Suspected Stroke: PHAST-TSC
Brief Title: Efficacy and Safety of Trans Sodium Crocetinate (TSC) for Treatment of Suspected Stroke
Acronym: PHAST-TSC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to lack of meaningful enrollment due to the COVID-19 pandemic.
Sponsor: Diffusion Pharmaceuticals Inc (Industry)
Collaborators: University of California, Los Angeles (Other); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100-501
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-12

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — trans-sodium crocetinate

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, placebo-controlled, double-blind, parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: TSC injections will be prepared and injected by unblinded personnel on each ambulance. All other study personnel will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trans Sodium Crocetinate (Experimental): Trans sodium crocetinate (TSC) will be administered intravenously as a bolus to subjects randomized to experimental drug. The bolus dose will consist of 0.25 mg/kg of TSC based on the estimated subject weight.
  Interventions: Drug: Trans-Sodium Crocetinate
- Placebo (Placebo Comparator): The placebo consists of commercially available sterile saline. Placebo will be administered intravenously as a bolus to subjects randomized to placebo. The volume of sterile saline will be based on the estimated subject weight.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Trans-Sodium Crocetinate — In the study drug kit containing the experimental drug (TSC), TSC will be reconstituted with the Sterile Water for Injection (USP) supplied in the same kit. There will be an unblinded paramedic who will reconstitute and inject the TSC on the ambulance.
  Other Names: TSC
  Arms: Trans Sodium Crocetinate
Other: Placebo — The study drug kit containing placebo (sterile saline for Injection) will be prepared and injected by the unblinded paramedic on the ambulance.
  Arms: Placebo

SUMMARY:
This study will assess the potential efficacy and safety of TSC as early treatment for both ischemic and hemorrhagic stroke when administered while subject is in ambulance being transported to hospital.

DETAILED DESCRIPTION:
This is a multicenter, randomized, placebo-controlled, double-blind, parallel group trial of intravenous trans sodium crocetinate (TSC) initiated by emergency medical service (EMS) responders in the field within 2 hours of symptom onset in 160 subjects with acute stroke. The primary objectives of the study are to evaluate the efficacy and safety of field-initiated TSC in improving the long-term functional outcome of subjects with acute stroke.

Subjects with acute stroke will be identified and screened in the ambulance by (EMS) responders who have received training in basic and advanced cardiac life support, stroke recognition, and specific procedures relevant to the proposed study. The EMS responders will contact a Study Neurologist, who will enroll eligible stroke patients into the study. Effort will be made to obtain prospective informed consent in the ambulance when deemed to be feasible. If not feasible, subjects will be enrolled under regulations for exception from explicit informed consent (EFIC) in emergency research circumstances, after public disclosure and community consultation. Written informed consent to continue in the study is obtained from subjects or their legally authorized representatives as soon as possible after hospital arrival.

EMS responders will deliver the single, field, bolus dose of study agent, TSC at 0.25 mg/kg or matched placebo, followed after hospital arrival by standard of care (SOC). No additional study drug will be administered in the hospital. Follow-up assessments will be performed at Emergency Department (ED) arrival, 24 hours, 48 hours, Day 4, Day 30, and Day 90. The study will be performed at up to 30 receiving hospital sites in Los Angeles County, CA, and central Virginia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-85, inclusive
2. Last known well time 15-120 minutes before anticipated study drug injection
3. Suspected stroke identified by the LAPSS
4. Moderate to severe motor deficit, with Los Angeles Motor Scale (LAMS) 2 or higher
5. No seizure

Exclusion Criteria:

1. Coma
2. Rapidly improving neurologic deficit
3. History of seizures or epilepsy
4. Pre-existing neurologic, psychiatric, or advanced systemic disease that would confound the neurological or functional outcome evaluations
5. SBP < 90 or > 220
6. Major head trauma in the last 24 hours
7. Recent stroke within 30 days
8. Known to be pregnant or lactating

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Southerland, MD, Principal Investigator — University of Virginia; Nerses Sanossian, MD, Principal Investigator — University of Southern California; Karen Johnston, MD, Study Chair — University of Virginia; Jeffrey Saver, MD, Study Chair — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Zachrison KS, Amati V, Schwamm LH, Yan Z, Nielsen V, Christie A, Reeves MJ, Sauser JP, Lomi A, Onnela JP. Influence of Hospital Characteristics on Hospital Transfer Destinations for Patients With Stroke. Circ Cardiovasc Qual Outcomes. 2022 May;15(5):e008269. doi: 10.1161/CIRCOUTCOMES.121.008269. Epub 2022 Apr 4. PMID 35369714

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trans Sodium Crocetinate | Placebo
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trans Sodium Crocetinate | Placebo | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Full Range); unit: years] | 74.0 [73 to 75] | 63.8 [45 to 80] | 67.2 [45 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Global Disability Level on the Modified Rankin Score (mRS)
Description: Modified Rankin Scale (mRS) is a measure of global disability. Total scale range is 0-6, with lower values indicating better outcomes.
  0 = No symptoms at all
  1. = No significant disability despite symptoms; able to carry out all usual duties and activities
  2. = Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. = Moderate disability; requiring some help, but able to walk without assistance
  4. = Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. = Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. = Dead
Time Frame: 90 days
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Trans Sodium Crocetinate | Placebo
Number analyzed (Participants) | 2 | 3
score on a scale | 2.5 [2 to 3] | 3.0 [0 to 3]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the start of study drug administration through the end of the Day 90 follow-up visit.
Arm/Group | Trans Sodium Crocetinate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/4
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/4
Other Adverse Events (participants affected / at risk) | 1/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trans Sodium Crocetinate (N=2) | Placebo (N=4)
Hemorrhagic Transformation of Infarct (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cerebral Edema (Nervous system disorders) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trans Sodium Crocetinate (N=2) | Placebo (N=4)
Hypochromic Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was early terminated after 6 subjects were enrolled due to logistical issues surrounding the COVID-19 pandemic. Due to this low enrollment number, the statistical plan outlined in the protocol was not utilized. Data listings and tables were instead created, which captured data on the 6 subjects in a descriptive manner. Therefore, no substantive conclusions could be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03763929/Prot_000.pdf